CLINICAL TRIAL: NCT06183281
Title: Integrating Nonpharmacologic Strategies for Pain With Inclusion, Respect, and Equity (INSPIRE): Tailored Digital Tools, Telehealth Coaching, and Primary Care Coordination
Brief Title: Integrating Nonpharmacologic Strategies for Pain With Inclusion, Respect, and Equity
Acronym: INSPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R33NS129050 (NIH); R61NS129050 (NIH); R33NS129050 (NIH)
Record Dates: First submitted 2023-08-13; First posted 2023-12-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain
Keywords: Non-malignant chronic pain; Digital health; Health coaching; Health equity; Cognitive therapy; Mindfulness; Movement
MeSH Terms: conditions — Chronic Pain | interventions — Mindfulness; Movement

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into intervention or enhanced usual care conditions
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The INSPIRE chronic pain management system has three primary components: 1) a patient facing smartphone app that collects and interprets a comprehensive intake and patient reported outcomes (PROs), provides health education, and a tailored, modular self-management program that includes cognitive-behavioral therapy (CBT), physical therapy (PT), and mindfulness-based interventions (MBI), 2) a weekly telehealth visit with a pain coach that uses the PRO data and module engagement measures to guide the visit, and 3) enhanced primary care coordination achieved through pain coaching notes and alerts integrated into the electronic health record (EHR).
  Interventions: Behavioral: CBT, Mindfulness, and Movement
- Control (No Intervention): Control participants will receive educational materials about chronic pain and full workbook with non-pharmacologic strategies.

INTERVENTIONS:
Behavioral: CBT, Mindfulness, and Movement — Blended CBT, mindfulness, and movement delivered through a mobile app and supported by a weekly telehealth pain management coach.
  Arms: Intervention

SUMMARY:
INSPIRE creates a trilingual mobile app and telehealth coaching program to promote non-pharmacologic strategies for pain management with Black, Chinese, and Latinx communities in the San Francisco Bay Area. Years 1-2 will develop the app and test it with a brief single arm pilot starting in Nov 2023. A full two arm randomized controlled trial (RCT) will being in early 2025 with changes in PEG scores as the primary outcome. Secondary outcomes include Helping to End Addiction Longterm (HEAL) common data elements.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or older
2. speak English, Spanish, or Cantonese
3. have a UCSF Health or SFHN PCP
4. be willing to use a smartphone (iOS or Android - either their own or one provided by the study)
5. have chronic, non-malignant pain for at least 3 months
6. be willing to participate in a 12 month patient-centered chronic pain management study where they will be randomized into one of two comparison arms

Exclusion Criteria:

* Severe mental illness or other condition preventing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain Intensity and Interference on the 11-point Pain, Enjoyment of Life, and General Activity Scale (PEG) | Baseline, 3mo, 6mo, 12mo
  The PEG Pain Screening Tool is a validated, self-reported 3-question survey assessing pain severity, the extent to which pain interferes with enjoyment of life, and the extent to which pain interferes with general activity. Possible scores for each question range from 0 (no pain, no interference) to 10 (worst possible pain, worst possible interference). The average of scores from the three questions yields the PEG score. Change = (PEG score at time point - PEG score at baseline)

SECONDARY OUTCOMES:
Change from Baseline in Physical Functioning on the 5-point PROMIS Physical Function Short Form 6b | Baseline, 3mo, 6mo, 12mo
  The PROMIS Physical Function Short Form 6b is a validated, self-reported 6-question survey assessing someone's ability to do household chores, to go up and down stairs at a normal pace, to go for a 15-minute walk, to run errands or shop, to do more than two hours of physical labor, and to do moderate work around the house. Possible scores for each question range from 1 (unable to do) to 5 (able to do without difficulty). Lower scores are indicative of lower levels of physical functioning. Change = (score at time point - score at baseline)
Change from Baseline in Sleep Disturbance and Sleep Duration on the 5-point PROMIS Sleep Disturbance Short Form 6a | Baseline, 3mo, 6mo, 12mo
  The PROMIS Sleep Disturbance Short Form 6a is a validated, self-reported 6-question survey assessing quality of sleep. Possible scores for each question range from 1 (very good) to 5 (very poor). A higher score indicates greater sleep disturbance. Change = (score at time point - score at baseline)
Change from Baseline in Fear and Anxiety about Pain on the 5-point Pain Catastrophizing Scale Short Form 6 | Baseline, 3mo, 6mo, 12mo
  The Pain Catastrophizing Scale Short Form 6 is a validated, self-reported 6-question survey assessing thoughts and feelings that someone may have about their pain. Possible scores for each question range from 0 (not at all, no catastrophizing thoughts and feelings) to 4 (all the time, constant catastrophizing thoughts and feelings). Change = (score at time point - score at baseline)
Change from Baseline in Self-reported Depressive Symptoms on the 4-point Patient Health Questionnaire - 9 (PHQ-9) | Baseline, 3mo, 6mo, 12mo
  The PHQ-9 is a validated, self-reported 9-question survey assessing common symptoms of depression. Possible scores for each question range from 0 (not at all) to 3 (nearly every day). A higher score indicates a higher likelihood of depression. Change = (score at time point - score at baseline)
Change from Baseline in Self-reported Anxiety Symptoms on the 4-point General Anxiety Scale (GAD-7) | Baseline, 3mo, 6mo, 12mo
  The GAD-7 is a validated, self-reported 7-question survey assessing common symptoms of anxiety. Possible scores for each question range from 0 (not at all) to 3 (nearly every day). A higher score indicates a higher likelihood of general anxiety. Change = (score at time point - score at baseline)
Change from Baseline in Overall Satisfaction with Treatment on the 7-point Patient Global Impression of Change (PGIC) | Baseline, 3mo, 6mo, 12mo
  The Patient Global Impression of Change (PGIC) is a validated, self-reported 1-question survey assessing how much a patient's pain has improved since the start of treatment. Possible scores range from 0 (very much improved) to 6 (very much worse). Change = (score at time point - score at baseline)
Change from Baseline in Self-reported Alcohol Use Disorder Symptoms on the 5-point Alcohol Use Disorder Identification Test (AUDIT) | Baseline, 3mo, 6mo, 12mo
  The Alcohol Use Disorder Identification Test (AUDIT) is a validated, self-reported 10-question survey assessing common symptoms of alcohol use disorder. Possible scores for each question range from 0 (never) to 4 (4 or more times per week). Scores for each question are added up. A score of 8 or higher is considered to indicate hazardous or harmful alcohol use. Change = (score at time point - score at baseline)
Change from Baseline in Drug Abuse Screening Test (DAST) Score | Baseline, 3mo, 6mo, 12mo
  The Drug Abuse Screening Test (DAST) is a validated, self-reported 10-question survey assessing risk of drug abuse. Each question is answered with a "yes" or a "no". Answers that indicate possible risk of drug abuse are given a score of 1, while answers that do not indicate possible risk of drug abuse are given a score of 0. The scores for each question are then added together. Change = (score at time point - score at baseline)
Change from Baseline in Internalized Stigma of Mental Illness on the 4-point Internalized Stigma of Mental Illness Inventory (ISMI) | Baseline, 3mo, 6mo, 12mo
  The Internalized Stigma of Mental Illness Inventory (ISMI) is a validated, self-reported 29-question survey assessing a patient's attitude, beliefs, and behaviors relating to their mental illness. Possible scores range from 1 (strongly disagree) to 4 (strongly agree). The scores for each question are added together. A higher score indicates greater internalized stigma of mental illness. Change = (score at time point - score at baseline)
Change from Baseline in Self-reported Social Isolation on the 5-point PROMIS Social Isolation Short Form 8a | Baseline, 3mo, 6mo, 12mo
  The PROMIS Social Isolation Short Form 8a is a validated, self-reported 8-question survey assessing a the extent to which someone feels isolated socially. Possible scores range from 1 (never) to 5 (always). The scores for each question are added together. A higher score indicates more severe isolation. Change = (score at time point - score at baseline)
Change from Baseline in Clinician Self-reported Attitudes, Beliefs, and Perspectives about Mental Illness on the 5-point Opening Minds Survey for Health Care Providers | Baseline, 3mo, 6mo, 12mo
  The Opening Minds Survey for Health Care Providers is a validated, self-reported 20-question survey assessing health care providers' attitudes, beliefs, and perspectives about mental illness. Possible responses to each question are "Strongly Disagree", "Disagree", "Neither Agree nor Disagree", "Agree", and "Strongly Agree". No numeric scores are assigned to responses. Changes in responses between each time point and baseline will be evaluated qualitatively.
Change from Baseline in Patient Self-reported Trust of their Healthcare Provider(s) on the 5-point PROMIS Healthcare Relationship Trust (HCR) Scale | Baseline, 3mo, 6mo, 12mo
  The Healthcare Relationship Trust Scale is a validated, self-reported 13-question survey assessing how a patient feels about their health care provider. Possible scores range from 0 (none of the time) to 4 (all of the time). The scores for each question are added together. A higher score indicates greater trust of the patient's health care provider. Change = (score at time point - score at baseline)
Change from Baseline in Self-reported Pain Self-Efficacy on the 7-point Pain Self-Efficacy Questionnaire - Two Item Short Form (PSEQ-2) | Baseline, 3mo, 6mo, 12mo
  The Pain Self-Efficacy Questionnaire Two Item Short Form (PSEQ-2) is a validated, self-reported 2-question survey assessing a patient's ability to live and work despite their pain. Possible scores range from 0 (not at all confident) to 6 (completely confident). The scores for each question are added together. A higher score indicates greater self-efficacy. Change = (score at time point - score at baseline)
Change from Baseline in Self-reported Psychological Inflexibility on the 7-point Psychological Inflexibility in Pain Scale | Baseline, 3mo, 6mo, 12mo
  The Psychological Inflexibility in Pain Scale is a validated, self-reported 12-question survey assessing how a patient accepts and adapts to a life with chronic pain. Possible scores range from 1 (never true) to 7 (always true). The scores for each question are added together. A higher score indicates greater psychological inflexibility in pain. Change = (score at time point - score at baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Satterfield, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco General Hospital, San Francisco, California
  - UCSF Adult Primary Care Mt. Zion Clinic, San Francisco, California

IPD SHARING:
Plan to Share IPD: No
This project is part of the Helping to End Addiction Longterm (HEAL) initiative and will use the data sharing platform required for that consortia.

REFERENCES:
- [Derived] Ristau J, Okobi A, Miller MJ, Cheng J, Deviren S, Schwarz EB, Fairchild T, Tsoh JY, Aguilera A, Zheng-Huang CJ, Satterfield JM. Integrating nonpharmacologic strategies for pain with Inclusion, Respect, and Equity (INSPIRE): a digital health study protocol for a pragmatic multisite randomized controlled trial. Trials. 2026 Jan 8;27(1):109. doi: 10.1186/s13063-025-09402-8. PMID 41507957